CLINICAL TRIAL: NCT03349151
Title: Postoperative Results of Early Versus On-demand Maternal Feeding After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Esra Ozbasli, Instructor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2017/4
Record Dates: First submitted 2017-11-14; First posted 2017-11-21 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Cesarean Delivery; Feeding Patterns; Patient Satisfaction; Postoperative Nausea and Vomiting
Keywords: Postoperative maternal feeding, cesarean section
MeSH Terms: conditions — Feeding Behavior; Patient Satisfaction; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Prospective randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early feeding (Active Comparator): This group will be served soft meal diet served on postoperative 2nd hour on return to the ward.
  Interventions: Behavioral: Early feeding
- On- demand feeding (Placebo Comparator): This group will be served soft meal diet served whenever they wanted to eat on return to the ward.
  Interventions: Behavioral: On- Demand feeding

INTERVENTIONS:
Behavioral: Early feeding — Feeding on postoperative 2nd hour on return to the ward
  Arms: Early feeding
Behavioral: On- Demand feeding — Feeding whenever the patient asks for on return to the ward
  Arms: On- demand feeding

SUMMARY:
To compare early versus on demand maternal feeding after cesarean delivery regarding gastrointestinal complaints and patient's satisfaction.

DETAILED DESCRIPTION:
Two hundred uncomplicated singleton term pregnancies who had caesarean section under regional anaesthesia will be included in our trial. Patients will be randomized to a soft food diet (honey, skimmed cheese, soup, mashed potatoe, pudding, grissini) served on postoperative 2nd hour or whenever they wanted to eat on return to the ward. Thirty minutes after they eat their meal, nausea, vomiting, ileus and distention will be questioned. Participants will be provided with the visual analogue scale (VAS), which will be presented with a statement explaining what was intended to measure. Patient satisfaction before discharge from hospital will be recorded by the patient by using a 100-mm VAS (0= minimum satisfaction, 100= maximum satisfaction). Time to first flatus passage and defecation will be recorded after the caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated singleton term pregnancy
* Planned or intrapartum uncomplicated cesarean section
* Cesarean section under regional anesthesia

Exclusion Criteria:

* General anesthesia
* History of bowel surgery
* Prenatal diagnosis of fetal anomaly
* Maternal disease
* Intraoperative or immediate postoperative major complications

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 262 (Actual)
Dates: Start 2017-11-19 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | On postoperative day 2 before they are discharged from the hospital.
  The primary outcome is patient satisfaction before discharge from hospital, measured using a scale called visual analogue scale (VAS). It is a 100-mm long scale with adjectival descriptions at both end positions. There will be a statement explaining what was intended to measure. Participants will be asked to mark the VAS on the second they of the surgery before they are discharged from the hospital. On this scale 0= lack of satisfaction from the timing of having their meal after the surgery 100= full satisfaction from the timing of their meal after the surgery.

SECONDARY OUTCOMES:
Postoperative passage of flatus and defecation | Postoperative day 0 to day 2.
  The participants will be asked to inform the nurse when they have their first passage of flatus and defecation.
Postoperative gastrointestinal complaints | Thirty minutes after the surgery
  Thirty minutes after the surgery the nurse will question the patients if they have a complaint of nausea, vomiting or abdominal distention.
Postoperative pain medication | Postoperative from day 0 to day 2
  After the surgery the need for pain medication will be followed. The name of the medicine, the time when the pain killer was used, the dosage of the medicine will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mete Gungor, MD, Prof., Study Director — Acibadem MAA University
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Sariyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis plan might be shared when the study is completed.

REFERENCES:
- [Background] Bisgaard T, Kehlet H. Early oral feeding after elective abdominal surgery--what are the issues? Nutrition. 2002 Nov-Dec;18(11-12):944-8. doi: 10.1016/s0899-9007(02)00990-5. PMID 12431715
- [Background] Mangesi L, Hofmeyr GJ. Early compared with delayed oral fluids and food after caesarean section. Cochrane Database Syst Rev. 2002;2002(3):CD003516. doi: 10.1002/14651858.CD003516. PMID 12137699
- [Background] Masood SN, Masood Y, Naim U, Masood MF. A randomized comparative trial of early initiation of oral maternal feeding versus conventional oral feeding after cesarean delivery. Int J Gynaecol Obstet. 2014 Aug;126(2):115-9. doi: 10.1016/j.ijgo.2014.02.023. Epub 2014 Apr 29. PMID 24856433
- [Background] Wrench IJ, Allison A, Galimberti A, Radley S, Wilson MJ. Introduction of enhanced recovery for elective caesarean section enabling next day discharge: a tertiary centre experience. Int J Obstet Anesth. 2015 May;24(2):124-30. doi: 10.1016/j.ijoa.2015.01.003. Epub 2015 Jan 14. PMID 25794417
- [Background] Kramer RL, Van Someren JK, Qualls CR, Curet LB. Postoperative management of cesarean patients: the effect of immediate feeding on the incidence of ileus. Obstet Gynecol. 1996 Jul;88(1):29-32. doi: 10.1016/0029-7844(96)00131-7. PMID 8684757